CLINICAL TRIAL: NCT06064864
Title: Efficacy and Safety of Formulation Switching Between Subcutaneous Infliximab and Intravenous Infliximab in Patients With Crohn's Disease
Brief Title: Efficacy and Safety of Formulation Switching Between SC Infliximab and IV Infliximab in Patients With CD
Acronym: CHAMELEON
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Asan Medical Center (Other)
Collaborators: Seoul National University Hospital (Other); Severance Hospital (Other); Kyung Hee University Hospital (Other); Kyungpook National University Hospital (Other); Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Byong Duk Ye, Professor, Asan Medical Center
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 20220644
Record Dates: First submitted 2023-09-10; First posted 2023-10-03 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: Crohn's Disease
Keywords: Crohn's disease; Infliximab; Biosimilar; Remsima; Subcutaneous; Intravenous
MeSH Terms: conditions — Crohn Disease | interventions — Infliximab

STUDY DESIGN:
Intervention Model Description: In this study, CD (Crohn's disease) patients who achieved clinical response at week 30 after to Remsima (CT-P13, a biosimilar of infliximab) SC (subcutaneous formulation) will be randomly (1:1) assigned to intravenous infliximab (Remsima) group (Arm 2) or to continued infliximab (Remsima) SC group (Arm 3). The primary endpoint of the study is the non-inferiority of Arm 3 compared with Arm 2 in terms of deep remission rate at week 54. Non-responder at week 30 will be allocated to Arm 1 (intravenous infliximab [Remsima] 10 mg/kg) and the secondary endpoint is the non-inferiority of Arm 3 compared with Arm 1 in terms of deep remission rate at week 54. Through this study, the investigators aim to provide the clinical evidence for selecting the most optimal formulation of infliximab according to therapeutic response among Korean patients with CD.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Non-response to SC infliximab at week 30 and switched to infliximab IV 10 mg/kg every 8 weeks (Experimental): Patients with moderately to severely active Crohn's disease will be given IV (intravenous) infliximab 5 mg/kg at week 0 and 2. Then, they will be treated with SC (subcutaneous) infliximab every 2 weeks from week 6. At week 30. patients will be allocated to one of 3 arms according to their response to SC infliximab.
  [Arm 1] Non-responders at week 30: Switched to infliximab IV 10 mg/kg every 8 weeks
  Interventions: Drug: Infliximab-Dyyb
- Response to SC infliximab at week 30 and then, switched to infliximab IV 5 mg/kg every 8 weeks (Experimental): Patients with moderately to severely active Crohn's disease will be given IV (intravenous) infliximab 5 mg/kg at week 0 and 2. Then, they will be treated with SC (subcutaneous) infliximab every 2 weeks from week 6. At week 30. patients will be allocated to one of 3 arms according to their response to SC infliximab.
  [Arm 2] Response to SC infliximab at week 30 and then, randomly allocated to infliximab IV 5 mg/kg every 8 weeks
  Interventions: Drug: Infliximab-Dyyb
- Response to SC infliximab at week 30 and then, continued infliximab SC 120 mg every 2 weeks (Active Comparator): Patients with moderately to severely active Crohn's disease will be given IV (intravenous) infliximab 5 mg/kg at week 0 and 2. Then, they will be treated with SC (subcutaneous) infliximab every 2 weeks from week 6. At week 30. patients will be allocated to one of 3 arms according to their response to SC infliximab.
  [Arm 3] Response to SC infliximab at week 30 and then, randomly allocated to infliximab SC 120 mg every 2 weeks
  Interventions: Drug: Infliximab-Dyyb

INTERVENTIONS:
Drug: Infliximab-Dyyb — Continued infliximab SC 120 mg every other week, if response to SC infliximab at week 30
  Other Names: Infliximab

SUMMARY:
The goal of this prospective, multicenter, open-label, randomized controlled, non-inferiority trial is to test efficacy and safety of formulation switching between subcutaneous (SC) infliximab and intravenous (IV) infliximab in patients with moderately to severely active Crohn's disease (CD). The primary endpoint of this study is deep remission at week 54. The main questions this study aims to answer are:

Question-1) Is maintenance therapy with SC infliximab (120mg every 2 weeks) non-inferior to IV infliximab (5mg/kg every 8 weeks) in terms of deep remission at week 54? Question-2) Is maintenance therapy with SC infliximab (120mg every 2 weeks) non-inferior to IV infliximab (10mg/kg every 8 weeks) in terms of deep remission at week 54?

DETAILED DESCRIPTION:
Remsima (CT-P13) is the first biosimilar of infliximab and its intravenous (IV) formulation has been used for patients with active Crohn's disease (CD).

Recently, subcutaneous (SC) formulation of Remsima (Remsima SC) was developed and approved by the Korean FDA (Food and Drug Administration). However, until now, besides a registration trial, real-life experiences of Remsima SC is still limited and the efficacy and safety of switching from SC to IV Remsima is still unknown.

In this study, patients with moderately to severely active CD who achieve clinical response to SC Remsima at week 30 (IV Remsima 5mg/kg at week 0 and 2, followed by SC Remsima 120mg every 2 weeks from week 6) will be randomly (1:1) assigned to IV Remsima group (Arm 2) or to continued SC Remsima group (Arm 3). Non-responders at week 30 will be allocated to Arm 1 (IV Remsima 10 mg/kg). The primary endpoint is the non-inferiority of Arm 3 compared with Arm 2 in terms of deep remission rate at week 54. The secondary endpoint is the non-inferiority of Arm 3 compared with Arm 1 in terms of deep remission rate at week 54. The non-inferiority margin is set as -20% and a total of 100 patients will be enrolled.

Through this study, the investigators aim to provide the clinical evidence for selecting the most optimal formulation of infliximab according to therapeutic response among Korean patients with CD.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years or older
2. Moderate to severe Crohn's disease (Crohn's disease activity index 220 to 450)
3. Ileocolonic Crohn's disease (CD) with Simple Endoscopic Score for Crohn Disease ≥6 or ileal or colonic CD with with Simple Endoscopic Score for Crohn Disease ≥4 and ulcer score ≥1 in at least one segment
4. Fecal calprotectin ≥250 µg/g or C-reactive protein≥0.5 mg/dL
5. Patients who have never been to exposed to any biologic agent
6. Patients who are non-responsive or intolerance to conventional therapy (corticosteroids, immunomodulators, or antibiotics, etc.) or contraindicated to conventional therapy
7. Patients who gave a voluntary informed consent

Exclusion Criteria:

1. Patients who have a history of hypersensitivity to humanized proteins
2. Patients ever treated with corticosteroids within 8 weeks of screening date
3. a) Symptomatic intestinal stricture, b) Symptomatic anal stricture, c) Untreated intra-abdominal abscess, d) Untreated perianal abscess, e) Abdominal surgery within 6 months, f) Patients who are expected to require intestinal surgeries during study period

   - However, the following patients can be included: from baseline, 4 weeks or more after proper drainage of perianal abscess and from baseline, 8 weeks or more after proper drainage of intra-abdominal abscess
4. Active tuberculosis. However, the following patients can be included: Patients who were diagnosed with tuberculosis, but were properly treated with anti-tuberculosis therapy according to the standard guidelines and who were confirmed to be cured.
5. Latent tuberculosis infection (LTBI): Patients confirmed as having latent tuberculosis through medical history, physical examination, chest X-ray, PPD (Purified Protein Derivative) skin test or interferon gamma release assay (IGRA) by a pulmonology specialist. However, patients with LTBI who finished proper treatment for LTBI for 4 weks and who are going to complete LTBI treatment.
6. HBsAg (Hepatitis B virus surface antigen)-positivity. Patients with negative HBsAg, but positive IgG anti-HBc (Immunoglobulin G anti-Hepatitis B core antibody) should be tested for HBV (hepatitis B virus) DNA real time quantitative PCR (polymerase chain reaction). If HBV DNA real time quantitative PCR ≥10 IU/mL should be excluded.
7. Anti-HCV (hepatitis C virus) antibody-positivity
8. History of HIV (human immunodeficiency virus) infection of positivity for anti-HIV
9. Heart disease of NYHA (New York Heart Association) Class III/IV
10. Active infection
11. Malignancy (excluding skin basal cell carcinoma, skin squamous cell carcinoma, and uterine cervix cancer) or history of colonic or small bowel dysplasia within 5 years
12. Pregnancy or lactating woman
13. Patients who are not applying proper contraceptive measures and patients who do not have a plan for proper contraceptive measures for at least 6 months after the last dose of infliximab (oral, parenteral, or implantable hormonal contraceptives, diaphragm, condom, intra-uterine device, or abstinence are accepted as proper contraceptive methods.
14. Patients who are decided to be not proper to be enrolled into the study by investigators.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-10-09 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Deep remission rate of Arm 3 compared with Arm 2 | Week 54
  Deep remission: all of these 3 criteria (1) CDAI (Crohn's disease activity index) <150, (2) SES-CD (Simple Endoscopic Score for Crohn's disease) ≤2, (3) No systemic corticosteroids use for at least 8 weeks before evaluation.
  CDAI can range from 0 to 600 and a higher value mean more clinically active disease.
  SES-CD is scored for 5 segments (ileum, right colon, transverse colon, left colon, and rectum) for (1) ulcer size, (2) % of ulcerated surface, (3) % of affected surface, and (4) the presence of stenosis. A higher value means a high endoscopic disease activity.
  The non-inferiority of Arm 3 compared with Arm 2 will be test and the non-inferiority margin will be set as "-20%".

SECONDARY OUTCOMES:
Deep remission rate of Arm 3 compared with Arm 1 | Week 54
  Deep remission: all of these 3 criteria (1) CDAI (Crohn's disease activity index)<150, (2) SES-CD (Simple Endoscopic Score for Crohn's disease) ≤2, (3) No systemic corticosteroids use for at least 8 weeks before evaluation.
  CDAI can range from 0 to 600 and a higher value mean more clinically active disease.
  SES-CD is scored for 5 segments (ileum, right colon, transverse colon, left colon, and rectum) for (1) ulcer size, (2) % of ulcerated surface, (3) % of affected surface, and (4) the presence of stenosis. A higher value means a high endoscopic disease activity.
  The non-inferiority of Arm 3 compared with Arm 1 will be test and the non-inferiority margin will be set as "-20%".
Corticosteroid-free endoscopic remission rate of each arm | Week 54
  All of these 2 criteria should be met to be classified as a corticosteroid-free endoscopic remitter: (1) SES-CD (Simple Endoscopic Score for Crohn's disease) ≤2, (2) No systemic corticosteroids use for at least 8 weeks before evaluation SES-CD is scored for 5 segments (ileum, right colon, transverse colon, left colon, and rectum) for (1) ulcer size, (2) % of ulcerated surface, (3) % of affected surface, and (4) the presence of stenosis. A higher value means a high endoscopic disease activity.
Corticosteroid-free complete mucosal healing rate of each arm | Week 54
  All of these 2 criteria should be met to be classified as an achiever of corticosteroid-free complete mucosal healing: (1) No visible ulcers (including aphthous ulcers) in ileocolonoscopy, (2) No systemic corticosteroids use for at least 8 weeks before evaluation
Corticosteroid-free clinical response (CDAI-70) rate of each arm | Week 54
  All of these 2 criteria should be met to be classified as a corticosteroid-free clinical responder (CDAI-70): (1) Reduction of CDAI (Crohn's disease activity index) 70 or more compared with the baseline, (2) No systemic corticosteroids use for at least 8 weeks before evaluation CDAI can range from 0 to 600 and a higher value mean more clinically active disease.
Corticosteroid-free clinical response (CDAI-100) rate of each arm | Week 54
  All of these 2 criteria should be met to be classified as a corticosteroid-free clinical responder (CDAI-100): (1) Reduction of CDAI (Crohn's disease activity index) 100 or more compared with the baseline, (2) No systemic corticosteroids use for at least 8 weeks before evaluation CDAI can range from 0 to 600 and a higher value mean more clinically active disease.
Corticosteroid-free clinical remission rate of each arm | Week 54
  All of these 2 criteria should be met to be classified as a corticosteroid-free clinical remitter: (1) CDAI (Crohn's disease activity index) < 150, (2) No systemic corticosteroids use for at least 8 weeks before evaluation CDAI can range from 0 to 600 and a higher value mean more clinically active disease.
Corticosteroid-free biochemical remission rate of each arm | Week 54
  All of these 2 criteria should be met to be classified as a biochemical remitter: (1) Both fecal calprotectin<250 µg/g and serum CRP (C-reactive protein) <0.5 mg/dL, (2) No systemic corticosteroids use for at least 8 weeks before evaluation
Rate of anti-drug antibody positivity in each arm | Week 54
  Proportion of patients with a positive anti-infliximab antibody compared with the baseline
The proportion of patients with treatment-related adverse events | Week 54
  Comparing the proportions of patients having any adverse events, serious adverse events, serious infections, and all types of adverse events as assessed by CTCAE v6.0

OTHER OUTCOMES:
Exploratory outcomes: trough level of infliximab to reach deep remission | Week 30
  Trough level of infliximab at week 30 (before infliximab administration) to reach deep remission at week 54
Exploratory outcomes: trough level of infliximab to reach clinical remission | Week 30
  Trough level of infliximab at week 30 (before infliximab administration) to reach clinical remission at week 54

CONTACTS AND LOCATIONS:
Overall Officials: Byong Duk Ye, MD, PhD, Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, South Korea

REFERENCES:
- [Background] Ye BD, Pesegova M, Alexeeva O, Osipenko M, Lahat A, Dorofeyev A, Fishman S, Levchenko O, Cheon JH, Scribano ML, Mateescu RB, Lee KM, Eun CS, Lee SJ, Lee SY, Kim H, Schreiber S, Fowler H, Cheung R, Kim YH. Efficacy and safety of biosimilar CT-P13 compared with originator infliximab in patients with active Crohn's disease: an international, randomised, double-blind, phase 3 non-inferiority study. Lancet. 2019 Apr 27;393(10182):1699-1707. doi: 10.1016/S0140-6736(18)32196-2. Epub 2019 Mar 28. PMID 30929895
- [Background] Schreiber S, Ben-Horin S, Leszczyszyn J, Dudkowiak R, Lahat A, Gawdis-Wojnarska B, Pukitis A, Horynski M, Farkas K, Kierkus J, Kowalski M, Lee SJ, Kim SH, Suh JH, Kim MR, Lee SG, Ye BD, Reinisch W. Randomized Controlled Trial: Subcutaneous vs Intravenous Infliximab CT-P13 Maintenance in Inflammatory Bowel Disease. Gastroenterology. 2021 Jun;160(7):2340-2353. doi: 10.1053/j.gastro.2021.02.068. Epub 2021 Mar 5. PMID 33676969
- [Background] Colombel JF, Rutgeerts PJ, Sandborn WJ, Yang M, Camez A, Pollack PF, Thakkar RB, Robinson AM, Chen N, Mulani PM, Chao J. Adalimumab induces deep remission in patients with Crohn's disease. Clin Gastroenterol Hepatol. 2014 Mar;12(3):414-22.e5. doi: 10.1016/j.cgh.2013.06.019. Epub 2013 Jul 12. PMID 23856361